CLINICAL TRIAL: NCT01905813
Title: A Phase 1, Open-label, Dose Escalation, Safety and Tolerability Study of INCB040093 in Subjects With Previously Treated B-Cell Malignancies
Brief Title: Study of INCB040093 in Subjects With Previously Treated B-Cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 40093-102
Record Dates: First submitted 2013-06-19; First posted 2013-07-23 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: B-cell Malignancies
MeSH Terms: interventions — itacitinib; INCB039110

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- INCB040093 (Experimental)
  Interventions: Drug: INCB040093
- INCB040093 in combination with itacitinib (INCB039110) (Experimental)
  Interventions: Drug: INCB040093 + itacitinib

INTERVENTIONS:
Drug: INCB040093 — Escalating doses starting at 100 mg every day (QD)
  Arms: INCB040093
Drug: INCB040093 + itacitinib — INCB040093 dose to be determined at completion of Part 1 of the study + itacitinib at a starting dose of 400 mg, QD with escalations planned up to 600 mg QD.
  Other Names: itacitinib (INCB039110)
  Arms: INCB040093 in combination with itacitinib (INCB039110)

SUMMARY:
The study will be conducted in three parts. Part 1 is a dose escalation phase to determine the maximum tolerated dose (MTD) of INCB040093, a PI3Kδ inhibitor, or a tolerated, pharmacologically active dose; Part 2 will evaluate the combination of INCB040093 and itacitinib (INCB039110), a JAK1 inhibitor, to determine the MTD of the combination or a tolerated dose that produces substantial pharmacologic inhibition of both targets; Part 3 will further evaluate the chosen doses of INCB040093 alone and in combination with itacitinib (INCB039110) in subjects with relapsed/refractory B-cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

• Aged 18 years or older, with lymphoid malignancies of B-cell origin as follows:

*Indolent / aggressive B-cell (NHL) Non- Hodgkin's Lymphoma:

EXCLUDING: Burkitt lymphoma and precursor B-lymphoblastic leukemia/lymphoma

INCLUDING: any non-Hodgkin's B-cell malignancy such as CLL and rare non-Hodgkin's B-cell subtypes such as Hairy Cell Leukemia, Waldenstrom macroglobulinemia, Mantle cell lymphoma, transformed NHL histologies, etc.

*Hodgkin's lymphoma

* Life expectancy of 12 weeks or longer.
* Subject must have received ≥ 1 prior treatment regimen.
* The subject must not be a candidate for potentially curative therapy, including stem cell transplant.

Exclusion Criteria:

* Received an investigational study drug within 28 days or 5 half-lives (whichever is longer) prior to receiving the first dose of study drug.
* Received any approved anticancer medications within 21 days or 5 half-lives (whichever is longer) prior to receiving their first dose of study drug (42 days for nitrosoureas) EXCEPT steroids at ≤ 10 mg prednisone daily (or equivalent).
* Has any unresolved toxicity ≥ Grade 2 from previous anticancer therapy.
* Has history of brain metastases or spinal cord compression, or lymphoma involving the central nervous system.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of ≥ 3.
* Received allogeneic hematopoietic stem cell transplant within the last 6 months, or has active graft versus host disease (GVHD) following allogeneic transplant, or is currently receiving immunosuppressive therapy following allogeneic transplant.
* Received autologous hematopoietic stem cell transplant within the last 3 months.
* Laboratory parameters not within the protocol-defined range.
* Current or recent history (<30 days prior to screening and/or <45 days prior to dosing) of a clinically meaningful bacterial, fungal, parasitic or mycobacterial infection.
* Current clinically active viral infection.
* Known history of infection with the human immunodeficiency virus (HIV).
* History of active hepatitis or positive serology for hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2013-06-30 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-04-17 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of INCB040093 as monotherapy and when given in combination with itacitinib as determined by clinical laboratory assessments, physical exams, 12-lead ECG and summary of adverse events | Measured every 3 weeks until progression.

SECONDARY OUTCOMES:
Preliminary efficacy as assessed by Overall Response Rate (ORR) as measured by published criteria for Hodgkin's/non-Hodgkin's lymphoma (Cheson et al 2007 and Owen et al 2013) and Chronic Lymphocytic Leukemia (CLL) (Cheson et el 2012) | Every 12 weeks (4 cycles) until study withdrawal
Pharmacokinetic (PK) collections. | Measured for each patient at Cycle 1 Day 1, Cycle 1 Day 8 and Cycle 1 Day 15
  Plasma concentrations of each INCB040093 and itacitinib will be used to estimate peak plasma concentration (Cmax) and area under the plasma concentration-time curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, MD, Study Director — Incyte Corporation
Locations (6):
- United States (6):
  - Birmingham, Alabama
  - Jacksonville, Florida
  - Ann Arbor, Michigan
  - Rochester, Minnesota
  - New York, New York
  - Rochester, New York

REFERENCES:
- [Derived] Phillips TJ, Forero-Torres A, Sher T, Diefenbach CS, Johnston P, Talpaz M, Pulini J, Zhou L, Scherle P, Chen X, Barr PM. Phase 1 study of the PI3Kdelta inhibitor INCB040093 +/- JAK1 inhibitor itacitinib in relapsed/refractory B-cell lymphoma. Blood. 2018 Jul 19;132(3):293-306. doi: 10.1182/blood-2017-10-812701. Epub 2018 Apr 25. PMID 29695516
- See also: Study of INCB040093 in Subjects With Previously Treated B-Cell Malignancies — https://incyteclinicaltrials.com/studies/incb-40093-102